CLINICAL TRIAL: NCT06991764
Title: Investigating the Effectiveness of a 2-week High-frequency Transcranial Pulsed-current Stimulation on Cognitive Outcomes in Healthy Adults: A Randomised, Double Blinded, Sham-controlled Study
Brief Title: Investigating the Effectiveness of a 2-week Novel Non-invasive Brain Stimulation Technique on Cognitive Outcomes in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Collaborators: Ministry of Education, Singapore (Other Government); National Institute of Education, Singapore (Other)
Responsible Party: Principal Investigator, Teo Wei Peng, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB-2025-003
Record Dates: First submitted 2025-04-11; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Transcranial Direct Current Stimulation (tDCS); Ageing; Executive Functioning; Transcranial Electric Stimulation
Keywords: Randomised Controlled Trial; Non-Invasive Brain Stimulation; Executive Functioning; Transcranial Direct Current Stimulation; Transcranial Pulsed Current Stimulation; Healthy Adults; Ageing
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to 1 of 3 conditions.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Transcranial Direct Current Stimulation (tDCS) (Active Comparator): In this condition, current intensity will be maintained between 0.6 to 0.7 mA for 20 minutes.
  Interventions: Device: Non-Invasive Brain Stimulation (tDCS / tPCS / sham-tPCS)
- High Frequency Transcranial Pulsed Current Stimulation (HF-tPCS) (Experimental): In this condition, current will be introduced in pulses with intensity consistent between 0.6 to 0.7 mA. The duration of the stimulation is 20 minutes.
  Interventions: Device: Non-Invasive Brain Stimulation (tDCS / tPCS / sham-tPCS)
- Sham-tPCS (Sham Comparator): In this condition, there will be a 30 seconds ramp-up phase to a current intensity between 0.6 to 0.7 mA followed by a 30 seconds ramp-down phase to 0 mA. The participant will, however, remain seated with the set-up for the remaining time until 20 minutes is up.
  Interventions: Device: Non-Invasive Brain Stimulation (tDCS / tPCS / sham-tPCS)

INTERVENTIONS:
Device: Non-Invasive Brain Stimulation (tDCS / tPCS / sham-tPCS) — This is a novel non-invasive brain stimulation technique that we hope to be investigating, and this technique will be compared with an active control (tDCS) and a control (sham-tPCS).

SUMMARY:
The goal of this randomised controlled trial is to investigate the effects of a 2-week high-frequency transcranial pulsed current stimulation (tPCS) on cognitive outcomes in older and healthy adults. The main questions it aims to answer are:

1. Would a single session of anodal tPCS over the left prefrontal cortex improve working memory, task inhibition, and task switching in healthy young and older adults, compared to anodal transcranial direct current stimulation (tDCS) and sham-tPCS?
2. Would repeated session of anodal-tPCS (2-weeks) lead to improvements in working memory, task inhibition, and task switching in healthy young and older adults, compared to tDCS and sham-tPCS?
3. Will tPCS be better tolerated among healthy adults, compared to tDCS?

Researchers will compare tPCS / tDCS / sham-tPCS to see if there are any differences in cognitive outcomes after 1 session and after repeated sessions, as well as to compare the tolerance of tPCS against tDCS and sham-tPCS.

Participants will be requested to:

* Undergo 1 of 3 of the following conditions: tDCS / tPCS / sham-tPCS
* Complete three sessions of cognitive tasks testing working memory, inhibition and task switching at baseline (pre-stimulation), after day 1 of brain stimulation and after 10 sessions of brain stimulation (post- repeated stimulation)
* Undergo fNIRS-EEG brain measurements concurrently with the cognitive tasks

DETAILED DESCRIPTION:
tPCS / tDCS and sham-tPCS will be administered between 0.6 to 0.7 mA for 20 minutes. This will take place over 10 consecutive sessions, with a 2 day break between days 5 and 6 of brain stimulation. The setup of the stimulation consists of a saline-soaked sponge anode electrode placed over the left forehead area over the left dorsal lateral prefrontal cortex, and the cathode will be placed over the right parietal cortex. Participants will be randomly assigned to 1 of 3 conditions and this will be blinded to both the participants and the researcher (double-blinded).

Cognitive tasks will be administered at baseline, after 1 session of stimulation and after 10 sessions of stimulation (post-stimulation). These cognitive tasks consist of a working memory task (1/2/3 back tasks), a cognitive inhibition task (go/no-go task) and a cognitive flexibility task (Stroop task). Concurrent with the cognitive task will be the administration of fNIRS-EEG recording to measure changes in brain activation and patterns during the tasks.

The experiment will take place in the Motor Behaviour Lab at the National Institute of Education, Nanyang Technological University in Singapore.

ELIGIBILITY:
Inclusion Criteria:

* Male and female young (21 to 30 years) and older adults (60 to 75 years)
* Right-handed
* Must be a native English speaker
* No clinical diagnosis of neurodevelopmental, mood, neurological or neurodegenerative disorders
* Adults with cardiometabolic or cardiovascular conditions may participate if their condition is controlled and stable with medication and / or lifestyle interventions

Exclusion Criteria:

* Currently on long-term medication for pain or migraines / headaches
* Adults with metallic implants in the chest or head region
* Adults with epilepsy, or known seizure or immediate family members that have had a seizure before
* Had a recent head injury that resulted in a temporary loss of consciousness or of memory in the last 12 months
* Had prior head surgery
* Prone to fainting
* Sensitive skin or prone to skin allergies

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Executive Functioning | Baseline, after day 1 of stimulation, 3 to 4 days after the 10 sessions of stimulation
  Working memory through 1-, 2- and 3-back tasks performance Behavioural inhibitory control through Go / No-Go task performance Cognitive flexibility through Stroop task performance
Task-based activation and functional connectivity during executive functioning tasks | Baseline, after day 1 of stimulation, 3 to 4 days after the 10 sessions of stimulation
  Measuring changes in hemodynamic (oxyhaemoglobin) responses in the brain using Functional Near-Infrared Spectroscopy (fNIRS)
Neural function associated with executive functioning tasks | Baseline, after day 1 of stimulation, 3 to 4 days after the 10 sessions of stimulation
  Measuring neural activity using electroencephaogram (EEG) whereby traditional EEG bands (e.g. Alpha, Beta, Theta, Delta) will be assessed.

SECONDARY OUTCOMES:
Tolerance of tPCS (intervention) | Immediately after the intervention
  Questionnaires on participants' well-being after stimulation sessions [adapted and modified from Antal et al. (2017)]. The participants will rate their symptoms / discomfort as follows: none, mild, moderate, or strong and state the extent to which the symptoms / discomfort is / are affecting their general state from a scale of 'Not at all' to 'Very much'.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Teo, Associate Professor, Principal Investigator — National Institute of Education, Nanyang Technological University, Singapore

IPD SHARING:
Plan to Share IPD: No